CLINICAL TRIAL: NCT01171365
Title: Small Particle Inhaled Steroids in Refractory Steroid-responsive Asthma
Brief Title: Small Particle Steroids in Refractory Asthma
Acronym: SPIRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09115
Record Dates: First submitted 2010-06-24; First posted 2010-07-28 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
Keywords: Ciclesonide; Asthma; Therapeutic Uses; Pulmonary Eosinophilia; Nitric Oxide; Lung Diseases; Respiratory Tract Diseases
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia; Lung Diseases; Respiratory Tract Diseases | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciclesonide (Active Comparator): Ciclesonide 320 microgrammes twice daily
  Interventions: Drug: Ciclesonide
- Placebo (Placebo Comparator): Placebo 2 inhalations twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide — Inhaled ciclesonide 320mcg twice daily
  Other Names: Alvesco
  Arms: Ciclesonide
Drug: Placebo — Matched placebo inhaler two inhalations twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether an inhaled steroid with a small particle size can be an additional treatment option in patients with refractory eosinophilic asthma.

DETAILED DESCRIPTION:
We have identified a group of patients with refractory asthma who have ongoing eosinophilic airway inflammation despite high dose inhaled corticosteroids.

Traditional inhaled steroids have a relatively proximal airway distribution which may lead to inadequate treatment of the distal airways.

We aim to demonstrate that a steroid inhaler with a smaller particle size which targets the distal airways can be a useful additional treatment option in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* ACQ >1.5 or a requirement for oral steroids twice a year or more
* High dose inhaled steroid (>1000mcg BDP or equivalent)
* Treatment with or unsuccessful trial of:

  * long-acting beta agonist
  * leukotriene antagonist
* Sputum eosinophil count >3% despite high dose inhaled steroid or >2% with serum eosinophils >0.4x10exp9/l
* Clinical response to 2 weeks of oral prednisolone: (any one)

  * reduction in ACQ by 0.5 or more
  * increase in FEV1 by 200ml
  * normalisation of exhaled nitric oxide or reduction of >25ppb

Exclusion Criteria:

* Current smoker, or ex-smoker for <12 months
* Current treatment with an extrafine steroid inhaler
* Respiratory infection within the last 4 weeks
* Pregnancy or lactation
* Poor compliance with usual asthma medication
* Clinical diagnosis of significant bronchiectasis
* Use of a medication which may interact with ciclesonide:

  * ketoconazole or itraconazole
  * ritonavir, nelfinavir

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in sputum eosinophil count over the trial period | 0 weeks (start), 8 weeks (finish)
  Sputum will be processed for a differential cell count, with the primary outcome the difference in sputum eosinophil count between active and placebo groups at 8 weeks

SECONDARY OUTCOMES:
Change in alveolar nitric oxide level over the trial period | 0 weeks (start), 4 weeks, 8 weeks (finish)
  alveolar nitric oxide has been shown to correlate with eosinophil count on BAL samples. Measured by measuring exhaled nitric oxide at multiple flow rates.
Change in bronchial nitric oxide level | 0 weeks (start), 4 weeks, 8 weeks (finish)
  Measured by single flow exhaled nitric oxide at 50 ml/s
Change in prebronchodilator FEV1 | 0 weeks (start), 4 weeks, 8 weeks (finish)
  Prebronchodilator FEV1 and FVC will be recorded with a Vitalograph Wedge Bellows spirometer
Change in Juniper Asthma Control Questionnaire (ACQ) score | 0 weeks (start), 4 weeks, 8 weeks (finish)
  UK English Version 2001
Change in Juniper Asthma Quality of Life Questionnaire (AQLQ) score | 0 weeks (start), 4 weeks, 8 weeks (finish)
  Self-administered United Kingdom Version 1994
Use of oral steroid over the trial period | 0-8 weeks
  Dose and duration of any additional oral corticosteroid will be documented
Number of patients with adverse events as a measure of safety and tolerability | 0-8 weeks
  Adverse events will be recorded throughout the trial period

CONTACTS AND LOCATIONS:
Overall Officials: Tim Harrison, Principal Investigator — University of Nottingham; Ian Pavord, Principal Investigator — University Hospitals, Leicester
Locations (2):
- United Kingdom (2):
  - University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire

REFERENCES:
- [Derived] Hodgson D, Anderson J, Reynolds C, Meakin G, Bailey H, Pavord I, Shaw D, Harrison T. A randomised controlled trial of small particle inhaled steroids in refractory eosinophilic asthma (SPIRA). Thorax. 2015 Jun;70(6):559-65. doi: 10.1136/thoraxjnl-2014-206481. Epub 2015 Apr 9. PMID 25858909